CLINICAL TRIAL: NCT06550661
Title: Effects of Ba Duan Jin on Muscle Strength, Balance, Cardiorespiratory Endurance, Body Composition and Quality of Life of Older People
Brief Title: Effects of Ba Duan Jin Training for Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chiu Shu-Ching, Assistant Professor, Central Taiwan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CTU112-SHOW-002
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Exercise; Old Age
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ba duan jin training (Experimental): twice a week
  Interventions: Behavioral: Ba duan jin
- usual care (No Intervention): once a week with video

INTERVENTIONS:
Behavioral: Ba duan jin — a kind of exercise
  Arms: Ba duan jin training

SUMMARY:
Baduanjin is one of the widely circulated fitness methods. The Ministry of Health, the Ministry of Education and the General Administration of Sports of China have vigorously promoted it as one of the contents of health and physical education classes, and promoted it as a health Qigong method throughout mainland China. It can be seen that Baduanjin's gentle and non-aggressive movements are suitable for physical training for people of all ages.

ELIGIBILITY:
Inclusion Criteria:

* (1) old person able to communicate and follow instructions, (2) stable and with sufficient physical strength: able to maintain at least one sitting position in a wheelchair or on the edge of a bed.

Exclusion Criteria:

* (1) Difficulty standing or walking and obvious musculoskeletal disease, (2) Diagnosed and recommended by a physician Those who are not suitable for sports activities, (3) serious diseases/unstable conditions, such as severe cardiopulmonary, liver and kidney diseases, severe malignant tumors, severe malnutrition, severe dementia, (4) more than 180 minutes of exercise per week in the past month time, (5) severe arrhythmia, (6) no intention to participate.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Chang in muscle strength from baseline to 12 weeks | Baseline and 12 weeks
  pinch, grip and quadriceps strength. A Higher score means a better outcome.
Chang in weight of muscle and fat from baseline to 12 weeks | Baseline and 12 weeks
  muscle mass(kg/%), fat mass (kg/%)
Chang in Activities of Daily Living from baseline to 12 weeks | Baseline and 12 weeks
  This is a scale of physical function. The range for total score is 0-100. A Higher score means a worse outcome.
Chang in Instrumental activities of daily living from baseline to 12 weeks | Baseline and 12 weeks
  This is a scale of physical function. The range for total score is 0-24. A Higher score means a better outcome.
Chang in short form Berg balance scale from baseline to 12 weeks | Baseline and 12 weeks
  Balance Assessment. The range is 0-4. A Higher score means a better outcome.
Chang in Gait analyses from wearable sensors from baseline to 12 weeks | Baseline and 12 weeks
  MTC mean magnitude and variability, as well as the stride-to-stride variability, stride time and length, lower limb peak angular velocity, and foot forward linear speed
Chang in EQ5D from baseline to 12 weeks | Baseline and 12 weeks
  This is a scale of quality of life. The range for total is 0-20. A higher score means a worse outcome.
Chang in WHOBREF from baseline to 12 weeks | Baseline and 12 weeks
  This is a scale of quality of life. A higher score means a better outcome.

SECONDARY OUTCOMES:
age, gender, married, religion, sleep, fall, disease status, education | Baseline
  Demographic basic data
height, weight | Baseline
  height(cm), weight(kg)
Clinical Dementia Rating | Baseline
  Mental Function Assessment. The range is 0-3. A Higher score means a worse outcome.
Chang in Cumulative Illness Rating Scale | Baseline
  A Higher score means a worse outcome. Range Min and Max to 0-56.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu, Principal Investigator — Central Taiwan University of Science and Technology
Locations (1):
- Show Chwan Memorial Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Chen CF, Chiu SC, Chiang CK, Lu YW. Effects of seated Baduanjin training modalities on body composition, muscle strength, and gait parameters in older adults: A cluster-randomised controlled trial. Complement Ther Med. 2025 Dec;95:103300. doi: 10.1016/j.ctim.2025.103300. Epub 2025 Nov 8. PMID 41213338